CLINICAL TRIAL: NCT04097613
Title: The Efficacy of Topical Povidone - Iodine Rinses in the Management of Biofilm-associated Chronic Rhinosinusitis
Brief Title: Betadine Rinses for Chronic Rhinosinusitis Prospective Cohort Study
Acronym: Betadine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Amin Javer, Clinical Professor, St. Paul's Hospital, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H17-01373
Record Dates: First submitted 2019-03-18; First posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
Keywords: Betadine; Povidone Iodine; CRS; Biofilm; Recalcitrant
MeSH Terms: conditions — Disease | interventions — Povidone-Iodine; Budesonide

STUDY DESIGN:
Intervention Model Description: Cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Betadine Treatment (Experimental): Study subjects will use betadine saline sinus rinse for period of 6 weeks.
  Interventions: Drug: Povidone-Iodine; Drug: Budesonide

INTERVENTIONS:
Drug: Povidone-Iodine — Povidone Iodine solution 5% (0.5% available iodine) by 3MTM has been specially formulated as a nasal antiseptic. They have shown topical application to be clinically safe, tolerable and to be rapidly bacteriocidal against aerobic gram positive and gram- negative bacteria including methicillin resistant Staphylococcus aureus, methicillin resistant Staphylococcus epidermidis, vancomycin resistant Enterococcus faecium and Enterococcus faecalis (VRE) and yeast (3M study 05-011100,05-011017, 05-011322).
  Other Names: Betadine
Drug: Budesonide — Budesonide is is provided in nebules (1mg/2cc). Patients will place two nebules of budesonide into the 250mls of saline.
  Other Names: Pulmicort

SUMMARY:
Povidone Iodine solution is a nasal antiseptic. Its application has been shown to be clinically safe, tolerable and effective against bacteria and fungi associated with chronic rhinosinusitis.

This study will evaluate the effectiveness of Povidone Iodine in this hard-to-treat patient group. Furthermore, the study will also further evaluate any side effects that may occur with the use of Povidone Iodine.

DETAILED DESCRIPTION:
Background and scientific rationale Chronic rhinosinusitis (CRS) is an inflammatory condition of the paranasal sinuses affecting millions of patients, resulting in billions of dollars being spent annually in associated health care costs. Biofilm has been implicated in chronic rhinosinusitis recalcitrant to appropriate medical therapy and well-executed endoscopic sinus surgery. The presence of biofilm results in patients having worse postoperative symptoms, recurrent infections, and persistent inflammation. Biofilms are bacterial or fungi communities surrounded by an extracellular polysaccharide matrix, which facilitates attachment to mucosa, survival, protection and proliferation. This configuration allows for resistance to innate host defenses and resistance to antibiotic therapy.

Povidone Iodine solution 5% (0.5% available iodine) by 3MTM has been specially formulated as a nasal antiseptic. They have shown topical application to be clinically safe, tolerable and to be rapidly bacteriocidal against aerobic gram positive and gram- negative bacteria including methicillin resistant Staphylococcus aureus, methicillin resistant Staphylococcus epidermidis, vancomycin resistant Enterococcus faecium and Enterococcus faecalis (VRE) and yeast(3M study 05-011100,05-011017, 05-011322).

Iodine is the active antimicrobial component in PVP-I. It has potent bactericidal, fungicidal and viricidal properties. It is an important element in the human body and is not known to be an allergen. Therefore there are no true allergies to iodine but rare cases of intolerance. In Japan, it is commonly recommended to gargle with PVP-Ito prevent upper respiratory infections. A prospective study evaluating the effect of mouth rinsing on iodine absorption and thyroid function showed that use of the mouthwash 4 times a day for 2 weeks or once a day for 24 weeks did not affect thyroid function. An evidence based review of randomized controlled trials and comparative studies determining the efficacy and risk associated with PVP-I irrigations used in general surgery, cardiovascular surgery, urological surgery, and orthopedic surgery found no significant risk were associated with the PVP-I irrigations other than increasing serum iodine.

There is a paucity of published data on the use of iodine during or after sinus surgery to treat biofilm. This study aims to determine if topical PVP-I rinses will result in an improvement in disease severity as determined by endoscopic scores (Modified Lund-Kennedy score). Secondly, as biofilm has been recognized as a source of poor outcomes in patients with recalcitrant chronic sinusitis (CRS), the study aims to determine if there's a significant reduction in biofilm biomass (bacterial or fungal) within the sinuses of recalcitrant CRS patients. In addition, the study will evaluate if there is a significant symptomatic improvement with the use of iodine rinses post-operatively.

Primary Objective:

To determine differences in Modified Lund-Kennedy (MLK) endoscopic score after 6 weeks of using Povidone-iodine (PVP-I) sinus rinses.

Secondary Objectives:

1. To determine if the use of Povidone iodine (PVP-I) sinus rinses reduces the number/density of biofilm colony forming units (bacterial or fungal) seen on mucosal biopsy of the sinus with evidence of recalcitrant/recurrent chronic rhinosinusitis (CRS) after 6 weeks.
2. To determine if the use of PVP-I sinus rinse improves disease specific quality of life in recalcitrant/recurrent CRS patients.

   Baseline Evaluation

   The following information will be obtained from each participant

   Demographic data:

   Age Gender Smoking status

   Clinical data:

   Thyroid function test (TSH and FT3/FT4 levels if indicated) at baseline and 6 weeks Eosinophil and Basophil levels Serum IgE levels Bacterial and fungal cultures (at baseline and 6weeks) History of sinus surgery Smell test at baseline and 6 weeks Saccharin test (Baseline and after 6 weeks)

   Conduct of the Study:

   Upon enrollment in the study, demographic data and clinical data will be obtained. The patient will be asked to fill out a SNOT-22 questionnaire, endoscopic pictures will be taken, culture taken via a suction trap and a biopsy of the sinus lining evidently affected by biofilm. The biopsy is painless and does not usually require local anesthesia but will be used if requested by the patient. A single bite of the mucosa is taken to remove tissue approximately 1x1mm. Bleeding is temporary and resolves spontaneously. Baseline smell test (University of Pennsylvania Smell Identification Test) followed by a saccharin test is done. All of the above except for the saccharin test and mucosal biopsy are a part of the routine clinical examination done for the patients in the rhinology clinic. A saccharin test will be used to establish the baseline cilia function, which is known to be denuded by biofilm13.

   The biopsy will be examined for biofilm (density and type of colony forming units) by scanning electron microscopy at the Centre for High-Throughput Phenogenomics at the University of British Columbia (UBC), part of the UBC Imaging Labs27.

   The patient will then be sent for baseline blood work (thyroid function test, IgE, eosinophil and basophil levels) and instructed to rinse with PVP-I added to their regular saline rinse. They will continue using the rinse for 6 weeks until they come back for their follow-up visit.

   Patients will then be seen 6 weeks later. They will be required to fill out the SNOT-22 questionnaire and would undergo endoscopic examination, smell and saccharin test. A biopsy is then taken from an adjacent site to the one taken upon enrollment in the study. They will then be sent for repeat eosinophil, basophil, IgE and TFTs levels. A blood test is a normal part of the evaluation done for the rhinology patient. The addition of the TFT will not require more injections for the patient.

   Management of Patient Care

   Patients have the right to withdraw from the study at any time. Patients who experience signs and symptoms of hypersensitivity to iodine, burning, itching, pain redness, tiredness, nausea or vomiting will be asked to stop the rinses immediately. The reaction will be noted and the code will be broken so that a discussion can occur between the physician and the patient regarding the use of iodine with the nasal rinses. Patients who meet any of the exclusion criteria that were not noted at the beginning of the study will be removed from this study and the physician will discuss the future management options with the patient.

   Drugs

   Povidone Iodine (PVP-I)

   Dosing and Administration

   PVP-I is provided in the form of a liquid at a concentration of 10% (1% available iodine). 2 mL of PVP-I will be diluted into 250 mL of saline solution. The final concentration of available iodine in the solution would be 0.008%.

   Dose Schedule:

   Patient will dilute 2 mL of 10% iodine into a 250 mL rinse bottle once a day

   Duration of therapy:

   The patient will administer the PVP-I or Saline rinse for 6 weeks

   Side effects

   The literature has some isolated reports of adverse reactions to iodine administration to include burning, swelling, and pain. No documented episode of anaphylaxis due to iodine has been identified in the literature. There are reports of TSH suppression with excessive mouth gargles with iodine, however, this is quickly reverses upon cessation of use.

   Budesonide

   Dosing and Administration:

   Budesonide is provided in nebules (1mg/2cc). Patients will place two nebules of budesonide into the 250mls of saline

   .

   Dose Schedule:

   Patients will administer the rinse once a day (2mg per day in total).

   Duration of Therapy:

   Patients will administer the budesonide for the entire duration of the study (42 days).

   Side Effects:

   Budesonide is generally well tolerated. The most common side-effect is drying of the nose, which may lead to nose bleeds.

   Inhaled budesonide may cause dysphonia, sore throat, and oralpharyngeal candidiasis. Headaches, asthenia and pain have been attributed to inhale budesonide as well. There are a number of ide effects which require consideration if topical budesonide reaches similar plasma concentrations as oralbudesonide, which include: depression, aggression, irritability, anxiety, psychosis, increased appetite, confusion, insomnia, nervousness, sleep disorder, amnesia, somnolence, reduction in bone density, chest pain, palpitations, tachycardia, dependent edema, facial edema, hypertension, flushing, increased C-reactive protein, acne, alopecia, dermatitis, eczema, increased sweating and skin disorders.

   Sample Size:

   Based on a retrospective study from our centre (St. Paul's Sinus Centre), that noted change in MLK score for 69 patients who used PVP-I, we were able to calculate a sample size for our prospective cohort study. 15 patients (30 sinus cavities) will be required to have an 80% chance at detecting a statistically significant (p-value < 0.05) decrease in MLK score. To account for a drop-out rate of 25% we plan to recruit 19 patients.

   Analysis:

   The primary outcome will be the change in MLK score before and after PVP-I use for 6 weeks. Secondary outcomes will be patient-reported quality of life (SNOT-22) and difference in biofilm CFUs. Descriptive statistics (mean, median, SD) will be used to describe demographic characteristics of the patients. The difference in MLK scores, CFUs, and SNOT-22 before and after treatment within and between groups will be analyzed using paired and unpaired students t-tests based on the variance of the outcomes.

   Safety Monitoring

   Patients who experience signs and symptoms of iodine reaction will be noted and the code will be broken so that a discussion can occur between the research supervisor and the patient regarding the use of the topical iodine.

   Patients can contact the office anytime if they notice any of the signs or symptoms of iodine reaction and will be seen by the research supervisor (or designate) within 24 hours.

   Adverse Events (AE's)

   All expected and unexpected adverse events will be recorded and graded by the research supervisor. Stablechronic conditions, which are present prior to the clinical trial entry and do not worsen, are not consideredadverse events and will be accounted for in the patient's medical history.

   Recording/Documentation of Adverse Events

   During each patient visit, the research supervisor will ask appropriate questions and perform a physical exam to elicit any adverse events. The research supervisor will also review blood work obtained from the patient. All reportable adverse events will be recorded on appropriate case report form. The research supervisor will also write the stop date, the severity of the AE and his judgment of the AE's relationship to the study.

   Serious Adverse Events (SAE's)

   An SAE is defined as an AE meeting one of the following:
   * Death occurring between Day 0 and 42 of the study.
   * Life Threatening Event (defined as a participant at immediate risk of death at the time of the event)
   * In-patient hospitalization or prolongation of existing hospitalization between Day 0 and 42 of the study.
   * Results in a persistent or significant disability/incapacity

   In the event of SAE, the research supervisor will discuss with the patient (or next of kin) whether there is a relationship between the study and the SAE. If there is a relationship, the PI will be responsible for coordinating care for the patient until the SAE has been addressed.

   Pregnancy During the Trial Patients will be responsible for determining if they are pregnant or become pregnant during the study. If patients notify the PI they are pregnant, they will be removed from the study and the medical management options will be discussed.

ELIGIBILITY:
Inclusion Criteria

* 19 years or older
* Diagnosed with CRS with biofilm recalcitrant/recurrent after a trial of at least 3 months of a combination of well executed sinus surgery, regular irrigation with topical steroids or mucosal atomization device and surfactants24
* Continued symptoms colored nasal discharge, post nasal drip, nasal congestion, decreased sense of smell, mucosal edema or polyps despite the above stated intervention

Exclusion Criteria

* Patients with sinonasal tumors.
* Patients with autoimmune diseases affecting the upper airway

  o eg Systemic lupus erythematosus, Sjögren's syndrome, systemic sclerosis etc.
* Immuno-compromised patients, and patients with impairment in mucociliary function

  o (e.g., cystic fibrosis, Kartagener syndrome)
* Hypersensitivity to iodine
* History of thyroid disorders including thyroid cancer, hyperthyroidism and hypothyroidism
* Use of medications for thyroid disorders including thyroxine and carbimazole
* Pregnancy
* Patients unable to speak English.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
MLK endoscopic grading | 6 weeks
  differences in Modified Lund-Kennedy (MLK) endoscopic score after 6 weeks of using Povidone-iodine (PVP-I) sinus rinses.

SECONDARY OUTCOMES:
Quality of Life determined by SNOT-22 Questionnaire | 6 weeks
  disease specific quality of life questionnaire score (SNOT-22) in recalcitrant/recurrent CRS patients

CONTACTS AND LOCATIONS:
Overall Officials: Amin Javer, M.D., Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
We will publish final outcomes as scientific paper.